CLINICAL TRIAL: NCT03545711
Title: Safety and Efficacy of Irinotecan Combined With Anlotinib in Patients With Pretreated Advanced Colorectal Cancer
Brief Title: Safety and Efficacy of Anlotinib in Combination With Irinotecan in Patients With Pretreated Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Huang, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC201803012
Record Dates: First submitted 2018-05-23; First posted 2018-06-04 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib plus Irinotecan (Experimental)
  Interventions: Drug: Anlotinib Hydrochloride with Irinotecan

INTERVENTIONS:
Drug: Anlotinib Hydrochloride with Irinotecan — Dose escalation of anlotinib starts from 8mg qd d1-14/q21d in combination with fixed dose of irinotecan at 180mg/m2 d1/q14d.

SUMMARY:
Patients with pretreated advanced colorectal cancer are recruited to the phase I portion of this prospective non-randomised study in an escalated dose cohort. The primary endpoint of the dose-escalation phase is to determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of anlotinib when given in combination with irinotecan. The phase II (dose-expansion) portion is designed to characterize the safety and potential efficacy of the combination therapy in pretreated advanced colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

* willing and able to provide written informed consent and comply with the requirements of the study
* histologically- or cytologically-confirmed advanced colorectal cancer
* failed or intolerable to at least one prior therapy
* have evidence of measurable disease per RECIST v1.1
* Eastern Collaborative Oncology Group (ECOG) Performance Status ≤ 1
* weight ≥40kg
* life expectancy >12 weeks

Exclusion Criteria:

Subjects meeting any of the following criteria are ineligible for participation in the study:

* history of any anti-cancer therapy (including investigational agents) within 28 days prior to study entry
* presence of toxicity of prior anti-cancer therapy that has not resolved to Grade 1, as determined by National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03
* symptomatic brain metastasis requiring active treatment
* any previous malignancy, except for non squamous-cell carcinoma of skin or carcinoma-in-situ of the uterine cervix within 5 years prior to study entry
* active or clinically unstable infection requiring systemic therapy
* unable to swallow oral medications or with gastrointestinal disorders that might interfere with proper absorption of oral drugs
* active digestive ulcer disease, inflammatory bowel disease, intestinal obstruction or any other condition that, in the clinical judgment of the Principal Investigator, may cause severe gastrointestinal bleeding or perforation
* unstable pulmonary embolism, deep vein thrombosis, or other significant arterial/venous thromboembolic event ≤2 months prior to study entry
* history of stroke or transient ischemic attack (TIA) within 12 months prior to study entry
* any of the following abnormal findings in organ or marrow function 1 week prior to study entry:

  * Leukocytes < 1.5*10^9/L, or Platelets < 100*10^9/L, or Hb< 90g/L
  * Total bilirubin > 1.5 × institutional upper limit of normal (ULN), or AST (aspartate amino transferase)/ALT (alanine amino transferase)> 3 × institutional ULN for liver metastases, > 1.5 × institutional ULN in case of no liver metastases
  * any electrolyte imbalance of clinical significance
  * creatinine > institutional ULN and creatinine clearance < 60 mL/min
  * spot urine protein ≥(2+) or 24-hour proteinuria ≥1.0g/24h
  * APTT (activated partial thromboplastin time) or INR (international normalized ratio for prothrombin time) > 1.5 × institutional ULN
* treatment refractory hypertension defined as a blood pressure of systolic> 140 millimeter of mercury (mm Hg) and/or diastolic > 90 mm Hg which cannot be controlled by a single anti-hypertensive agent
* LVEF (left ventricular ejection fraction ) <50%
* history of acute coronary syndromes (including myocardial infarction and unstable angina), coronary artery bypass graft within 6 months prior to study entry, or history or evidence of current ≥ Class II congestive heart failure as defined by New York Heart Association (NYHA)
* present with non-healing fractures of bone or wounds of skin
* pregnant or lactating female
* sexually active female (of childbearing potential) or male unwilling to adopt an effective method of birth control during the course of the study
* serious and/or unstable pre-existing psychiatric disorder
* familial, sociological or geographical conditions that, in the clinical judgment of the Principal Investigator, do not permit compliance with the protocol
* known immediate or delayed hypersensitivity reaction to anlotinib, irinotecan or their excipients
* administration of irinotecan in prior treatments

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-05-26 (Actual); Primary Completion 2019-11-24 (Estimated); Study Completion 2020-11-24 (Estimated)

PRIMARY OUTCOMES:
MTD | 6 months
  the maximum tolerated dose (MTD) of Anlotinib when administered in combination with fixed dose of irinotecan in advanced colorectal cancer patients.
ORR | 18 months
  the overall response rate (ORR) of Anlotinib when administered in combination with fixed dose of irinotecan in advanced colorectal cancer patients.

SECONDARY OUTCOMES:
DCR | 18 months
  the disease control rate (DCR) of the combination of Anlotinib with Irinotecan in pretreated advanced colorectal cancer patients.
PFS | 18 months
  the progression free survival (PFS) of the combination of Anlotinib with Irinotecan in pretreated advanced colorectal cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, MD, Principal Investigator — Cancer Hospital,CAMS
Locations (1):
- Jing Huang, Beijing, China

IPD SHARING:
Plan to Share IPD: No